CLINICAL TRIAL: NCT04422275
Title: Coronavirus Smell Therapy for Anosmia Recovery
Acronym: Co-STAR
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding not received
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jay F. Piccirillo, MD, Prof of Otolaryngology, Washington University School of Medicine
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PA-18-334
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Anosmia
Keywords: COVID; Smell Therapy
MeSH Terms: conditions — Anosmia | interventions — Budesonide

STUDY DESIGN:
Intervention Model Description: 2 x 2 factorial design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Budesonide & High-Concentration OLF (Active Comparator): In this arm, subjects will perform nasal saline lavage (240 ml) with budesonide (0.5mg/capsule) and four different high-concentration (1 ml) essential oils for olfactory training twice daily.
  Interventions: Drug: Budesonide; Behavioral: High-Concentration Essential Oil
- Placebo & High-Concentration OLF (Active Comparator): In this arm, subjects will perform nasal saline lavage (240 ml) with placebo (lactose monohydrate) and four different high-concentration (1 ml) essential oils for olfactory training twice daily.
  Interventions: Behavioral: High-Concentration Essential Oil; Drug: Placebo
- Budesonide & Low-Concentration OLF (Active Comparator): In this arm, subjects will perform nasal saline lavage (240 ml) with budesonide (0.5mg/capsule) and four different low-concentration (0.1 ml) essential oils for olfactory training twice daily.
  Interventions: Drug: Budesonide; Behavioral: Low-Concentration Essential Oil
- Placebo & Low-Concentration OLF (Placebo Comparator): In this arm, subjects will perform nasal saline lavage (240 ml) with placebo (lactose monohydrate) and four different low-concentration (0.1 ml) essential oils for olfactory training twice daily.
  Interventions: Drug: Placebo; Behavioral: Low-Concentration Essential Oil

INTERVENTIONS:
Drug: Budesonide — The drug intervention budesonide (0.5 mg /capsule) will be dissolved in 240 ml nasal saline lavage.
  Arms: Budesonide & High-Concentration OLF; Budesonide & Low-Concentration OLF
Behavioral: High-Concentration Essential Oil — High-concentration essential oil will include 1 ml of essential oil per jar.
  Arms: Budesonide & High-Concentration OLF; Placebo & High-Concentration OLF
Drug: Placebo — The placebo (lactose monohydrate) drug will be dissolved in 240 ml of nasal saline lavage.
  Arms: Placebo & High-Concentration OLF; Placebo & Low-Concentration OLF
Behavioral: Low-Concentration Essential Oil — Low-concentration essential oil will include 0.1 ml of essential oil per jar.
  Arms: Budesonide & Low-Concentration OLF; Placebo & Low-Concentration OLF

SUMMARY:
As the COVID-19 pandemic spread around the world, anosmia and dysgeusia were quickly recognized as two of the key presenting symptoms. The probability of return of smell is related to severity of smell loss at presentation, but it appears that the loss of sense of smell and taste seems to persist in approximately 10% of the affected patients after 6 months. As a result of COVID-19, it is estimated that within the next 12 months > 150,000 Americans will suffer permanent loss of smell. The magnitude of this impairment on the health, safety, and quality of life is truly unprecedented and makes post-COVID olfactory disorder a major public health problem. Thus, there is a pressing need to identify effective treatments.

The research questions are to determine the effects of steroid nasal saline lavage and olfactory training among adults with post-COVID olfactory dysfunction and identify confounders and modifiers of any observed effects. To answer the research question, the investigators propose a 2 x 2 factorial design blinded randomized clinical trial whereby 220 subjects with documented COVID-19 with anosmia/hyposmia of 12 weeks duration or longer from Missouri, Illinois, and Indiana will be recruited electronically from COVID patient advocacy sites, social media sites, and other internet sources. Enrolled subjects will be randomized to nasal saline lavage with topical budesonide or placebo to address the presumed role of inflammation in the olfactory cleft and each subject will also be randomized to olfactory training with patient-specific, high- or low-concentration essential oil scent to assess the role of olfactory training. Data will be analyzed in a blinded fashion to allow estimation of observed effect size for both anti-inflammatory and olfactory training.

This innovative study will exploit the unique opportunities presented by COVID-19. The study will use a high-tech virtual "contactless" research strategy, including eConsent and digital mHealth techniques to obtain rapid answers to the research questions. The interventions are low-cost, readily available, and results of this study can be directly disseminated to the care of COVID-19 patients with anosmia.

DETAILED DESCRIPTION:
This will be a virtual or "contactless" clinical trial. Subjects will be recruited through a variety of ways and will complete all baseline and post-intervention assessments via specially designed electronic platforms, including REDCap and digital eHealth assessments. There will be no in-person, on-campus interaction between the members of the study team and research participants.

Convalescent COVID-19 subjects with persistent (i.e. > 3 months) decreased sense of smell, and a score on the UPSIT consistent with decreased olfactory function (< 35 women, < 34 men) will be offered enrollment. This will be a 2 x 2 factorial double-blinded, placebo-controlled, randomized clinical trial.

Subjects will be assigned to one of two nasal saline lavage interventions through a randomization schedule developed by the Study Pharmacist. The package and detailed instructions will be shipped directly to the subject from pharmacy. Subjects will be requested to rinse each nasal cavity once daily for 12 weeks and to keep track of their daily use through a paper dairy or specially created app to track compliance.

Subjects will be assigned to one of two olfactory training interventions through a randomization schedule prepared by the Study Pharmacist. The smell training intervention will be shipped directly to the subject. The subject will be expected to complete the smell training for 12 weeks as instructed. Subjects will be asked to record their daily training on a specially created app and make observations on their smell or taste function at the end of every week.

Outcome assessments will be performed immediately upon completing nasal saline lavage and olfactory training (Week 12) and follow-up (Week 24).

ELIGIBILITY:
Inclusion Criteria:

* Adult women and men.
* Positive laboratory finding for SARS-CoV-2 (e.g., real-time reverse-transcription polymerase chain reaction (rRT-PCR) assays to detect viral RNA).
* In convalescence from their COVID-19 illness.
* Subjective complaints of reduced olfaction after COVID-19 infection of greater than 3 months duration.
* Reduced olfaction ability as determined by a score of <35 (women) or <34 (men) on the University of Pennsylvania Smell Identification Test (UPSIT ).
* Ability to read, write, and understand English.

Exclusion Criteria:

* History of olfaction disorder prior to COVID-19 infection.
* History of nasal cavity polyps.
* Dependence on prolonged corticosteroid therapy for comorbid conditions, such as asthma and chronic obstructive pulmonary disease.
* History of cerebrospinal fluid leak.
* History of allergy to budesonide or other topical steroids.
* Pregnant or breast feeding or intend to become pregnant during the course of the trial.
* Current infection or history of one of the following infections: Tuberculosis (TB) lung infection, or Herpes infection of the eye.
* Baseline UPSIT score 5 or below, which suggests malingering.
* History of neurodegenerative disease (i.e. Alzheimer's dementia, Parkinson's disease, Lewy body dementia, frontotemporal dementia).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
University of Pennsylvania Smell Identification Test (UPSIT) | The within subject change in UPSIT between baseline and 12- and 24-week assessment time frame.
  The University of Pennsylvania Smell Identification Test (UPSIT) (Sensonics, New Jersey)7 is the most widely accepted olfactory identification test in North America. The UPSIT consists of four 10-page booklets, with a total of 40 items. Subjects are asked to scratch each strip with a pencil to release the scents, detect the smell, and identify the smell from the four choice options. The UPSIT comes from a scoring rubric that identifies the normalcy benchmark based on age and gender. Normosmia is defined as ≥34 for males and ≥35 for females, and an increase of 4 points or more from baseline indicates a clinically meaningful improvement. UPSIT has high internal reliability across a wide range of populations.

SECONDARY OUTCOMES:
Questionnaire of Olfactory Disorders-Negative Statements (QOD-NS). | The within subject change in QOD-NS between baseline and assessment time frame.
  The Questionnaire of Olfactory Disorders-Negative Statements (QOD-NS) was adapted from the original 52-item Questionnaire of Olfactory Disorders. This short-modified version is a validated 17-item questionnaire about quality of life and impairments related to olfactory dysfunction. The maximum score is 51, and higher values indicate worse quality of life or higher degree of impairment of normal daily activity. Mean scores in anosmics is 19; hyposmics is 8; and normosmics is 0. Prior studies used a cutoff score of 12.5 to reflect normal vs. abnormal scores.The minimum clinically important difference is 5.2.
Global Rating of Smell. | 12 weeks - End of nasal lavage & olfactory training; 24 weeks - Follow-up (12 weeks after completion of lavage & training)
  The Global Rating of Smell is a single-item, global rating that asks:
  "Overall, please rate your current sense of smell? Excellent, Very Good, Good, Fair, Poor, Absent."
Global Rating of Smell Change. | 12 weeks - End of olfactory training; 24 weeks - Follow-up (12 weeks after completion of lavage & training)
  The Global Rating of Smell Change is a single-item, global rating that asks: "Compared to your sense of smell # weeks ago, how would you rate your change in smell since then? Much better, Somewhat better, Slightly better, Neither better nor worse, Slightly worse, Somewhat worse, or Much worse." The time frame ("#") will be changed to reflect the correct time since enrollment (i.e., 12, or 24 weeks).

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No